CLINICAL TRIAL: NCT05421832
Title: A Novel Measurement Concept to Objectively Quantify Severity of Vocal and Speech Related Symptoms Associated With Parkinson's Disease
Acronym: Voice-PD
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Koneksa Health (Industry); Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Tanya Simuni, MD, Professor, Northwestern University
Other Study IDs: STU00216902
Record Dates: First submitted 2022-06-08; First posted 2022-06-16 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- PD Cohort 1: PD patients assessed via the Hoehn & Yahr (H&Y) Scale to be in Stages 1-2 of PD (inclusive)
  Interventions: Device: Digital Speech Application
- PD Cohort 2: PD patients assessed via the H&Y Scale to be in Stages 3-4 of PD (inclusive)
  Interventions: Device: Digital Speech Application
- Prodromal PD: Patients who meet PI-defined criteria for prodromal PD, i.e., the latent phase of disease progression during which clinical PD symptoms have yet to manifest
  Interventions: Device: Digital Speech Application
- Age and Sex-matched Healthy Control: Age & sex matched healthy control subjects who have not been diagnosed with PD
  Interventions: Device: Digital Speech Application

INTERVENTIONS:
Device: Digital Speech Application — A custom smartphone-based speech assessment tool to extract multiple hypothesis-driven acoustic features from patient speech in a real-life environment.

SUMMARY:
The aim of this research program is to develop and validate a smartphone app-based digital measurement concept that:

* Objectively quantifies the severity of Parkinson's Disease (PD) related vocal and speech symptoms;
* Accurately and sensitively identifies vocal and speech abnormalities associated with the prodromal stage of PD.

DETAILED DESCRIPTION:
Although multiple approaches to this problem have been proposed in addition to commercially available speech analytics platforms, there is currently no established measure which incorporates the disparate aspects of affected speech to fully characterize Parkinson's symptom progression, particularly in the prodromal phase.

The measurement concept being evaluated in the present study utilizes a custom smartphone-based speech assessment tool to extract multiple hypothesis-driven acoustic features from patient speech in a real-life environment. The resultant features will be used to train a pair of supervised machine learning models to predict clinical PD symptom severity scores, and to distinguish prodromal PD patients from both healthy matched controls and PD patients in more advanced phases of disease progression.

ELIGIBILITY:
Inclusion Criteria:

PD:

1. Male or female age 30 years or older at Screening Visit.
2. Diagnosis of PD as defined by MDS PD diagnostic criteria [1]
3. PD severity at Screening Visit of either:

   * PD Hoehn and Yahr Stage 1-2, inclusive (PD Cohort I)
   * PD Hoehn and Yahr Stages 3-4, inclusive (PD Cohort II)
4. Able and willing to complete all aspects of the study, including at home smartphone app and Zoom telehealth assessments.
5. Able to provide informed consent.

Prodromal PD:

1. Confirmation that participant is eligible based on clinician determined predictive criteria of known risk of PD including

   1. Rapid eye movement sleep behavior disorder (RBD), possible, probable or definite, OR
   2. Hyposmia defined as less than 10th percentile on University of Pennsylvania Smell Identification Test (UPSIT), age and gender adjusted, OR
   3. Known genetic variants associated with PD risk, AND Confirmed eligible DAT scan.
2. Male or female age 30 or older at Screening Visit.
3. Able and willing to complete all aspects of the study, including at home smartphone app and Zoom telehealth assessments
4. Able to provide informed consent.

Age & Sex Matched Healthy Control:

1. Male or female age 30 years or older at Screening visit.
2. Able and willing to complete all aspects of the study, including at home smartphone app and Zoom telehealth assessments
3. Able to provide informed consent.

Exclusion Criteria:

PD:

1. Late-stage PD diagnosis (i.e., Hoehn & Yahr Stage 5) at Screening Visit
2. Symptomatic or atypical PD syndromes due to either drugs (e.g., metoclopramide, flunarizine, neuroleptics) or metabolic disorders (e.g., Wilson's disease), encephalitis, or degenerative diseases (e.g., progressive supranuclear palsy).
3. Current or active clinically significant neurological disorder other than PD (in the opinion of the Investigator).
4. Significant cognitive impairment or clinical dementia at Screening that, in the opinion of the Investigator, would interfere with study evaluation.
5. History of drug and/or alcohol abuse within the past year prior to Screening Visit.
6. Inability or unwillingness to complete all aspects of the study - including use of a provisioned smartphone for study assessments; completion of telehealth assessments.
7. Any other medical or psychiatric condition, which in the opinion of the investigator might preclude participation.

Prodromal PD:

1. Clinical diagnosis of PD, other parkinsonism, or dementia.
2. Any current or active clinically significant neurological disorder (in the opinion of the Investigator).
3. Previously obtained MRI scan with evidence of clinically significant neurological disorder (in the opinion of the Investigator).
4. Significant cognitive impairment or clinical dementia at Screening that, in the opinion of the Investigator, would interfere with study evaluation.
5. History of drug and/or alcohol abuse within the past year prior to Screening Visit.
6. Inability or unwillingness to complete all aspects of the study - including use of a provisioned smartphone for study assessments; completion of telehealth assessments.
7. Any other medical or psychiatric condition, which in the opinion of the investigator might preclude participation.

Age & Sex Matched Healthy Control:

1. First degree relative with PD (i.e., biologic parent, sibling, child).
2. Any current or active clinically significant neurological disorder (in the opinion of the Investigator).
3. Previously obtained MRI scan with evidence of clinically significant neurological disorder (in the opinion of the Investigator).
4. Significant cognitive impairment or clinical dementia at Screening that, in the opinion of the Investigator, would interfere with study evaluation.
5. History of drug and/or alcohol abuse within the past year prior to Screening Visit.
6. Inability or unwillingness to complete all aspects of the study - including use of a provisioned smartphone for study assessments; completion of telehealth assessments.
7. Any other medical or psychiatric condition, which in the opinion of the investigator might preclude participation

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * PD Cohort I (n=30): PD patients assessed via the Hoehn & Yahr (H&Y) Scale to be in Stages 1-2 of PD (inclusive)
  * PD Cohort II (n = 30): PD patients assessed via the H&Y Scale to be in Stages 3-4 of PD (inclusive)
  * Prodromal PD Cohort (n = 30): Patients who meet PI-defined criteria for prodromal PD, i.e., the latent phase of disease progression during which clinical PD symptoms have yet to manifest
  * Age & Sex Matched Healthy Control Cohort (n = 30) - age & sex matched healthy control subjects who have not been diagnosed with PD
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Compliance of digital speech assessment data recorded via smartphone assessments | 8 weeks
  o % Interpretable minutes of data per patient
Quality of digital speech assessment data recorded via smartphone assessments | 8 weeks
  o % Interpretable vs. expected number of minutes of data per patient by complete days on study
Usability of digital speech assessments | 8 weeks
  o SUS Usability scores by score, grade and adjective rating
Content validity of digital speech assessments | 8 weeks
  o Percent of patients that score Excellent or Good for usability ratings

SECONDARY OUTCOMES:
Characterization and reliability of digital speech assessment features | 8 weeks
  o Candidate feature characterization: response distributions, and outlier analysis. Stratification of sustained phonation measures by MDS-UPDRS relevant speech items
Reliability of digital speech assessment features | 8 weeks
  internal consistency and test-retest reliability
Predictive performance of machine learning (ML) regression model | 8 weeks
  o Construct validity: convergent validity of each model output versus relevant MDS-UPDRS speech items and Parts I-IV total score, respectively; and versus Hoehn & Yahr Stage
Predictive performance of ML classification model | 8 weeks
  o Known group validity by cohort (including by H&Y Stage/ MDS-UPDRS Parts I-IV total score)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No